CLINICAL TRIAL: NCT01773798
Title: A Trial Investigating the Pharmacodynamic and Pharmacokinetic Properties of Insulin Degludec/Insulin Aspart 15 in Subjects With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN1050-4008; 2012-004215-31 (EudraCT Number); U1111-1134-6222 (Other: WHO)
Record Dates: First submitted 2013-01-18; First posted 2013-01-23 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — insulin degludec; insulin degludec, insulin aspart drug combination; Insulin Aspart

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- IDegAsp 15 (Experimental)
  Interventions: Drug: insulin degludec/insulin aspart 15; Drug: placebo
- IDegAsp (Experimental)
  Interventions: Drug: insulin degludec/insulin aspart; Drug: placebo
- IDeg (Experimental)
  Interventions: Drug: insulin degludec
- IAsp (Active Comparator)
  Interventions: Drug: insulin aspart
- IDeg + IAsp (Experimental)
  Interventions: Drug: insulin degludec; Drug: insulin aspart

INTERVENTIONS:
Drug: insulin degludec/insulin aspart 15 — Each subject subject will be randomly allocated to five single doses. Administered subcutaneously (s.c, under the skin) on five dosing visits separated by 15-25 days. The dose level will be 0.5 U/kg Body Weight (BW).
  Arms: IDegAsp 15
Drug: insulin degludec/insulin aspart — Each subject subject will be randomly allocated to five single doses. Administered subcutaneously (s.c, under the skin) on five dosing visits separated by 15-25 days. The dose level will be 0.5 U/kg Body Weight (BW).
  Other Names: IDegAsp
  Arms: IDegAsp
Drug: insulin degludec — Each subject subject will be randomly allocated to five single doses. Administered subcutaneously (s.c, under the skin) on five dosing visits separated by 15-25 days. The dose level will be 0.425 U/kg Body Weight (BW).
  Arms: IDeg; IDeg + IAsp
Drug: insulin aspart — Each subject subject will be randomly allocated to five single doses. Administered subcutaneously (s.c, under the skin) on five dosing visits separated by 15-25 days. The dose level will be 0.075 U/kg Body Weight (BW).
  Arms: IAsp; IDeg + IAsp
Drug: placebo — Each subject subject will be randomly allocated to five single doses. Administered subcutaneously (s.c, under the skin) on five dosing visits separated by 15-25 days.
  Arms: IDegAsp; IDegAsp 15

SUMMARY:
This trial is conducted in Europe. The aim of the trial is to investigate the pharmacodynamic (the effect of the investigated drug on the body) and the pharmacokinetic (exposure of the trial drug in the body) properties of insulin degludec/insulin aspart 15 in subjects with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus (as diagnosed clinically) for at least 12 months
* Body mass index 18.0-28.0 kg/m^2 (both inclusive)

Exclusion Criteria:

* Subject who has donated any blood or plasma in the past month or more than 500 mL within 3 months prior to screening
* Smoker (defined as a subject who is smoking more than 5 cigarettes or the equivalent per day)
* Not able or willing to refrain from smoking, use of nicotine substitute products or transdermal nicotine patches during the inpatient period
* Female of childbearing potential who is pregnant, breast-feeding or intend to become pregnant or is not using adequate contraceptive methods (adequate contraceptive measures include sterilisation, hormonal intrauterine devices, oral contraceptives, condom with spermizide, sexual abstinence or vasectomised partner)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2013-01; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Area under the glucose infusion rate curve | From 0 to 6 hours after single dose (IDegAsp 15, IDeg and IDegAsp)

SECONDARY OUTCOMES:
Area under the serum IDeg concentration-time curve | From 0 to 120 hours after single dose
Area under the serum IAsp concentration-time curve | From 0 to 12 hours after single dose

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Graz, Austria

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com